CLINICAL TRIAL: NCT00089219
Title: Vaccination With Multiple Synthetic Melanoma Peptides Recognized by Helper T-Cells in Patients With Advanced Melanoma
Brief Title: Vaccine Therapy in Treating Patients With Stage IIIB, Stage IIIC, or Stage IV Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Craig L Slingluff, Jr, Professor of Surgery, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10464; UVACC-MEL-41; UVACC-28502
Record Dates: First submitted 2004-08-04; First posted 2004-08-05 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Intraocular Melanoma; Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma; ciliary body and choroid melanoma, medium/large size; extraocular extension melanoma; iris melanoma; recurrent intraocular melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — incomplete Freund's adjuvant; montanide ISA 51; Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A. 6MHP vaccine 200 mcg (Experimental): vaccine containing 6 melanoma helper peptides, at 200 mcg per peptide, with GM-CSF and IFA (Montanide ISA-51)
  Interventions: Biological: IFA; Biological: 6MHP; Biological: GM-CSF
- Arm B. 6MHP vaccine 400 mcg (Experimental): vaccine containing 6 melanoma helper peptides, at 400 mcg per peptide, with GM-CSF and IFA (Montanide ISA-51)
  Interventions: Biological: IFA; Biological: 6MHP; Biological: GM-CSF
- Arm C. 6MHP vaccine 800 mcg (Experimental): vaccine containing 6 melanoma helper peptides, at 800 mcg per peptide, with GM-CSF and IFA (Montanide ISA-51)
  Interventions: Biological: IFA; Biological: 6MHP; Biological: GM-CSF

INTERVENTIONS:
Biological: IFA — vaccine adjuvant
  Other Names: incomplete Freund's adjuvant, Montanide ISA-51
Biological: 6MHP — melanoma helper peptides
  Other Names: multi-epitope melanoma peptide vaccine
Biological: GM-CSF — vaccine adjuvant
  Other Names: sargramostim

SUMMARY:
RATIONALE: Vaccines may make the body build an immune response to kill tumor cells.

PURPOSE: This randomized phase I/II trial is studying three different doses of a vaccine and comparing them to see how well they work in treating patients with stage IIIB, stage IIIC, or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the immune response in patients with stage IIIB, IIIC, or IV melanoma treated with vaccine comprising multiple synthetic melanoma peptides, Montanide ISA-51, and sargramostim (GM-CSF).

OUTLINE: This is a randomized study. Patients are randomized to 1 of 3 treatment arms.

* Arm I: Patients receive vaccine comprising low-dose multiple synthetic melanoma peptides, Montanide ISA-51, and sargramostim (GM-CSF) on days 1, 8, 15, 29, 36, and 43.
* Arm II: Patients receive vaccine comprising medium-dose multiple synthetic melanoma peptides, Montanide ISA-51, and GM-CSF as in arm I.
* Arm III: Patients receive vaccine comprising high-dose multiple synthetic melanoma peptides, Montanide ISA-51, and GM-CSF as in arm I.

On day 22, the lymph node draining the vaccination site is removed to determine whether the immune system is responding to the vaccine.

PROJECTED ACCRUAL: A maximum of 38 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of stage IIIB, IIIC, or IV melanoma
* HLA-DR1, -DR4, -DR11, -DR13, or -DR15 positive
* Brain metastases allowed at the discretion of the principle investigator

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-1

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3
* Platelet count > 100,000/mm ^3
* Hemoglobin > 9 g/dL

Hepatic

* Liver function tests ≤ 2.5 times upper limit of normal (ULN)

Renal

* Creatinine ≤ 1.5 times ULN

Cardiovascular

* No New York Heart Association class III or IV heart disease

Other

* Prior diagnosis of other cancer allowed
* Not pregnant or nursing
* Weight ≥ 110 pounds
* No uncontrolled diabetes

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior growth factors
* More than 4 weeks since prior allergy shots
* More than 12 weeks since prior melanoma vaccine therapy* NOTE: *Prior melanoma vaccine allowed only for patients with disease progression during or after administration of the vaccine
* No prior vaccination with any of the peptides used in this study

Chemotherapy

* More than 4 weeks since prior chemotherapy

Endocrine therapy

* More than 4 weeks since prior steroids

Radiotherapy

* More than 4 weeks since prior radiotherapy

Surgery

* Not specified

Other

* More than 1 month since prior investigational drugs or therapies
* No other concurrent investigational drugs or therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2003-07; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Safety: Dose-limiting toxicity | During study period
  Toxicities measured by CTCAE.
Immunogenicity | day 22
  Melanoma peptide-specific helper T cell responses in the sentinel immunized node (SIN) on day 22.

SECONDARY OUTCOMES:
Immune response in the blood | day 50
  Immune response measured in the blood, by proliferation assay, over time during the study.
DTH response | by day 85
  Delayed-type hypersensitivity response to tumor peptides
Clinical outcome | during the study
  Clinical tumor response

CONTACTS AND LOCATIONS:
Overall Officials: Craig L. Slingluff, MD, Study Chair — University of Virginia
Locations (1):
- University of Virginia Cancer Center, Charlottesville, Virginia, United States

REFERENCES:
- [Result] Slingluff CL Jr, Petroni GR, Olson W, Czarkowski A, Grosh WW, Smolkin M, Chianese-Bullock KA, Neese PY, Deacon DH, Nail C, Merrill P, Fink R, Patterson JW, Rehm PK. Helper T-cell responses and clinical activity of a melanoma vaccine with multiple peptides from MAGE and melanocytic differentiation antigens. J Clin Oncol. 2008 Oct 20;26(30):4973-80. doi: 10.1200/JCO.2008.17.3161. Epub 2008 Sep 22. PMID 18809608
- [Derived] Shukla GS, Olson WC, Pero SC, Sun YJ, Carman CL, Slingluff CL Jr, Krag DN. Vaccine-draining lymph nodes of cancer patients for generating anti-cancer antibodies. J Transl Med. 2017 Aug 29;15(1):180. doi: 10.1186/s12967-017-1283-8. PMID 28851380
- [Derived] Dillon PM, Olson WC, Czarkowski A, Petroni GR, Smolkin M, Grosh WW, Chianese-Bullock KA, Deacon DH, Slingluff CL Jr. A melanoma helper peptide vaccine increases Th1 cytokine production by leukocytes in peripheral blood and immunized lymph nodes. J Immunother Cancer. 2014 Jul 15;2:23. doi: 10.1186/2051-1426-2-23. eCollection 2014. PMID 25126421